CLINICAL TRIAL: NCT06117696
Title: Optimizing the Announcement of Advanced or Metastatic Prostate Cancer Using Animated Videos (CartDiag PROSTATE)
Acronym: CartDiagPROST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PPRC12; 2023-A00446-39 (Other: IDRCB)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer advanced or metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Standard announcement system
- video reinforced announcment group: standard announcement system reinforced by animated videos
  Interventions: Other: Animated video

INTERVENTIONS:
Other: Animated video — delivery of written and oral information, supported by animated videos.
  Groups: video reinforced announcment group

SUMMARY:
In hospitals, the standard prostate cancer announcement system is based on oral and written information. To improve this system, we have developed animated videos that retrace the patient's care path.

This is an exploratory, controlled, before-and-after, multicenter study designed to assess the effect of a standard announcement system reinforced by animated videos on patients' level of understanding of prostate cancer diagnosis and treatment. Patients' perception of information will be assessed using the EORTC QLQ-INFO25 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Collection of the patient's non-opposition prior to participation in the study.
2. Patient aged ≥ 18 years at inclusion.
3. Patient with newly diagnosed advanced or metastatic prostate cancer.
4. Patients due to start systemic therapy.
5. Patients undergoing consultation.
6. Patient affiliated to a social security scheme.
7. Patient capable, according to the physician-investigator, of communicating well, understanding and complying with the requirements of the study.
8. Patient with a smartphone or computer to review the video at home.

Exclusion Criteria:

1. Patient related to any member of the study staff or having a close relationship or conflict of interest with the sponsor.
2. Patient to receive only local treatment.
3. Patient who does not understand French.
4. Clinical follow-up impossible for psychological, family, social or geographical reasons.
5. Vulnerable patient: deprived of liberty by judicial or administrative decision, adult subject to legal protection or unable to express non-opposition.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Study Population: Patient with newly diagnosed advanced or metastatic prostate cancer
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-INFO25 score | Through study completion (30 days)
  overall score of the EORTC QLQ-INFO25 questionnaire at D0 and D30 completed by the patient in each group

SECONDARY OUTCOMES:
EORTC QLQ-INFO25 score differences | Through study completion (30 days)
  difference in EORTC QLQ-INFO25 global score between D0 and D30 in each group

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - Clinique Hartmann, Neuilly-sur-Seine
  - HIA Bégin, Saint-Mandé
- CHU Pointe-à-Pître, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No